CLINICAL TRIAL: NCT04905264
Title: TIRESIA Project - Severe Acquired Brain Injuries: Prognostic Factors and Quality of Care
Brief Title: Severe Acquired Brain Injuries: Prognostic Factors and Quality of Care
Status: Recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: TIRESIA
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Brain Injuries, Acute
Keywords: Rehabilitation; Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults admitted in participating Rehabilitation Units for Severe Acquired Brain Injuries: Adults admitted in study's participants Rehabilitation Units for Severe Acquired Brain Injuries from the 1st of July 2021 to the 31st of December 2023. Patients entered into these units more than 14 weeks after the acute event are excluded

SUMMARY:
The main purpose of this project is to identify the medium-term prognostic factors for patients with Severe Acquired Brain Injuries and evaluate their impact.

The secondary aim is to create a system of continuous assessment of the quality of care for each rehabilitation unit.

DETAILED DESCRIPTION:
For each unit involved, it will be collected these data :

* Structural and organizational data of the Rehabilitation Units for Severe Acquired Brain Injuries;
* Detailed information on patients upon entering Rehabilitation Units for Severe Acquired Brain Injuries;
* Detailed information on patients, re-evaluated 4 months after the acute event

Statistical models will be implemented, in order to identify prognostic factors that could predict the probability to observe three events, which represent objectives of the rehabilitation process: decannulation, trunk control and total feeding by os. These events should be evaluated four months after the acute episode.

ELIGIBILITY:
Inclusion Criteria:

* patients with Serious Acquired Brain Injuries
* admission to rehabilitation units

Exclusion Criteria:

- patients admitted more than 14 weeks after the acute event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the Rehabilitation Units for Severe Acquired Brain Injuries participating in the study during the 30 months of enrollment provided by the research
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Tracheostomy tube | july 2021 - june 2025
  Removal of the tracheostomy tube, which is considered successful if the patient is not to be re-cannulated within 7 days
Trunk control | july 2021 - june 2025
  Achievement of trunk control, for which the patient must be able to maintain the sitting position for at least 60 seconds, on a rigid surface, with the lower limbs in support, but without support from the upper limbs and without rear support of the trunk
Total feeeding by os | july 2021 - june 2025
  Oral feeding with sufficient caloric intake

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bertolini, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (27):
- Italy (27):
  - Ospedale SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Centro di Riabilitazione Terranuova Bracciolini, Arezzo
  - Ospedale civile di Baggiovara, Baggiovara
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale Maggiore, Bologna
  - Fondazione Poliambulanza, Brescia
  - Ospedale S. Michele, AO Brotzu, Cagliari
  - Ospedale S. Sebastiano, Correggio
  - Istituto S. Anna, Crotone
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Fondazione Don Gnocchi, Florence
  - Ospedale di Foligno, Foligno
  - Montecatone Rehabilitation Institute SpA, Imola
  - USL Toscana Nord Ovest, Lucca
  - IRCCS S. Maria Nascente, Fondazione don Gnocchi, Milan
  - Istituto Palazzolo, Don Gnocchi, Milan
  - Ospedale Sacro Cuore don Calabria, Negrar
  - ATS Sardegna, Oristano
  - Ospedale Buccheri La Ferla Fatebenefratelli, Palermo
  - Centro Cardinal Ferrari, Parma
  - AUSL Piacenza, Piacenza
  - Centro di riabilitazione E. Spalenza, Don Gnocchi, Rovato
  - Ospedale "Casa Sollievo della Sofferenza", San Giovanni Rotondo
  - Fondazione Don Gnocchi, Sant'Angelo dei Lombardi, Sant'Angelo dei Lombardi
  - IRCCS Telese, ICS Maugeri, Telese Terme
  - Ospedale Riabilitativo Villa Rosa, Trento
  - A.ULSS n.8 Berica, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided
Protecting the privacy policy, all the data that underlie results in a publication will be shared. The scientific commettee of the study has to decide the criteria and the best way to share them

REFERENCES:
- [Derived] Nattino G, Acler M, Bargellesi S, Bertagnoni G, Carrara G, De Tanti A, Estraneo A, Ghilardi GI, Lavezzi S, Lombardi F, Lucca LF, Mancuso M, Montis A, Mule C, Navarro J, Posteraro F, Rossato E, Simoncini L, Bertolini G. A prospective multicenter study on prognostic factors and quality of care in Severe Acquired Brain Injury rehabilitation units: a project from the Tiresia network. Front Neurol. 2025 Feb 19;16:1527533. doi: 10.3389/fneur.2025.1527533. eCollection 2025. PMID 40046674